CLINICAL TRIAL: NCT04924816
Title: Evaluation of the Response to the Awake Prone Position in Patients With COVID-19
Brief Title: Awake Prone Position in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Brazilian Institute of Higher Education of Censa (Other)
Responsible Party: Principal Investigator, Luciano Matos Chicayban, Laboratório de Pesquisa em Fisioterapia Pneumofuncional e Intensiva (LAPEFIPI), Brazilian Institute of Higher Education of Censa
Other Study IDs: ISECENSA
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Awake prone position — The prone position in awake patients consists of asking the patient to voluntarily change to prone position, in a swimmer's posture

SUMMARY:
Although prone position is widely used in awake patients with COVID-19 associated with supplemental oxygenation, high flow nasal catheter, or noninvasive ventilation, few studies are attesting to its real benefits on physiological variables or intubation rate. Awake patients dependent on supplemental oxygen may have different responses to PP about peripheral oxygen saturation, heart rate, and respiratory rate. Such responses may be permanent, transient, or even absent. We believe that the response to PP can be a predictor of the need for admission to the ICU. This study aimed to evaluate the acute effects of different types of response to the prone position in patients awake with COVID-19.

ELIGIBILITY:
Inclusion Criteria: patients with a confirmed diagnosis of COVID-19, through tests based on PCR and chest tomography with suggestive findings, spontaneously ventilating, dependent on supplemental oxygen. The study included patients with: (1) age ≥ 18 years, (2) peripheral oxygen saturation less than 92% under supplemental oxygen administration equal to or greater than 6 L / min through a nasal catheter or reservoir mask; (3) no use of NIV or high-flow nasal catheter; (4) continuous monitoring with pulse oximeter; (5) mental status that allowed to follow the instructions; and (6) able to tolerate PP with minimal assistance.

-

Exclusion Criteria:

* hemodynamic instability, severe obesity, or who were unable to tolerate and cooperate with the performance of PP

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of COVID-19, spontaneously ventilating, dependent on supplemental oxygen.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
ICU admission rate | Patients were followed up for up to 15 days of hospitalization.
  The criteria defined for admission to the ICU included maintenance of SpO2 below 90% with oxygen flow at 15 L / min, RF greater than 30 incursions per minute, reduced level of consciousness, or clinical signs of persistent increase in respiratory work, such as paradoxical ventilatory pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Luciano M Chicayban, Campos dos Goytacazes, Rio de Janeiro, Brazil